CLINICAL TRIAL: NCT05936892
Title: Comparative Effects of UE Aerobic and Resistance Training on Cardiorespiratory Fitness in Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0309
Record Dates: First submitted 2023-06-14; First posted 2023-07-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Blood Pressure
Keywords: Cardiorespiratory Fitness; Oxygen Consumption

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- upper extremity aerobic training (Experimental): upper extremity aerobic training
  Interventions: Other: upper extremity aerobic training
- upper extremity resistance training (Experimental): upper extremity resistance training
  Interventions: Other: upper extremity resistance training

INTERVENTIONS:
Other: upper extremity aerobic training — upper extremity aerobic training & baseline treatment will be given. Overall session time will be 40-45 minutes
  Arms: upper extremity aerobic training
Other: upper extremity resistance training — upper extremity resistance training Overall session time will be 40-45 minutes
  Arms: upper extremity resistance training

SUMMARY:
simple random sampling into group A & group B to collect data. Group A will be given upper extremity aerobic training and group B will be given upper extremity resistance training. The study will be completed within the time duration of ten months. Primary Outcome measures of the research will be pain, range of motion, and quality of life.

DETAILED DESCRIPTION:
A randomized clinical trial will be conducted at Multan institute of cardiology, Multan. Non probability convenient sampling technique will be applied on--patients who will be allocated through simple random sampling into group A & group B to collect data. Group A will be given upper extremity aerobic training and group B will be given upper extremity resistance training. The study will be completed within the time duration of ten months. Primary Outcome measures of the research will be pain, range of motion, and quality of life. Data will be analyzed using SPSS software version 25. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age group of 35-65years
* Both male and females
* Patients with blood pressure >140/90mm Hg

Exclusion Criteria:

* Regular engagement in physical exercise training in past 4 weeks
* Patients with secondary hypertension
* Patients using more than one hypertensive drugs
* Recent myocardial infarction
* Congestive heart failure
* Uncontrolled cardiac arrythmia

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
6 MWT RESISTANCE TRAINING ON CARDIORESPIRATORY FITNESS IN HYPERTENSIVE PATIENTS | 4 weeks
  The 6MWT is a practical simple test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians. This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes (the 6MWD).The self-paced 6MWT assesses the submaximal level of functional capacity. (19) According to studies, the distance walked by a healthy subject on six-minute walk test ranges from 400 to 700m.
  * Men ranged from 735m to 580m.
  * Women ranged from 657m to 500m.

SECONDARY OUTCOMES:
Borg rating of perceived exertion (RPE) | 4 weeks
  Borg rating of perceived exertion (RPE) is an outcome measure scale used in knowing exercise intensity prescription. It is used in monitoring progress and mode of exercise in cardiac patients as well as in other patient populations undergoing rehabilitation and endurance training.Borg RPE scale was developed by Gunnar Borg for rating exertion and breathlessness during physical activity ; that is, how hard the activity is as shown by high heart and respiration rate , profuse perspiration and muscle exertion.
  RPE scale contains 10 points (20).
  * 1 denotes very light activity
  * 2-3 denotes light activity
  * 4-6 denotes moderate activity
  * 7-8 denotes vigorous activity
  * 9 denotes very hard activity
  * 10 denotes maximum effort activity training.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Faisal, MS.CPPT, Principal Investigator — Riphah International University
Locations (1):
- Multan Institute of Cardiology, Multan, Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kokubo Y. Prevention of hypertension and cardiovascular diseases: a comparison of lifestyle factors in Westerners and East Asians. Hypertension. 2014 Apr;63(4):655-60. doi: 10.1161/HYPERTENSIONAHA.113.00543. Epub 2014 Jan 13. No abstract available. PMID 24420548
- [Background] Franco OH, Peeters A, Bonneux L, de Laet C. Blood pressure in adulthood and life expectancy with cardiovascular disease in men and women: life course analysis. Hypertension. 2005 Aug;46(2):280-6. doi: 10.1161/01.HYP.0000173433.67426.9b. Epub 2005 Jun 27. PMID 15983235
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; ESC Scientific Document Group. 2018 ESC/ESH Guidelines for the management of arterial hypertension. Eur Heart J. 2018 Sep 1;39(33):3021-3104. doi: 10.1093/eurheartj/ehy339. No abstract available. PMID 30165516
- [Background] Smart TFF, Doleman B, Hatt J, Paul M, Toft S, Lund JN, Phillips BE. The role of resistance exercise training for improving cardiorespiratory fitness in healthy older adults: a systematic review and meta-analysis. Age Ageing. 2022 Jun 1;51(6):afac143. doi: 10.1093/ageing/afac143. PMID 35737600
- [Background] Mandsager K, Harb S, Cremer P, Phelan D, Nissen SE, Jaber W. Association of Cardiorespiratory Fitness With Long-term Mortality Among Adults Undergoing Exercise Treadmill Testing. JAMA Netw Open. 2018 Oct 5;1(6):e183605. doi: 10.1001/jamanetworkopen.2018.3605. PMID 30646252
- [Background] Khalid Z, Farheen H, Tariq MI, Amjad I. Effectiveness of resistance interval training versus aerobic interval training on peak oxygen uptake in patients with myocardial infarction. J Pak Med Assoc. 2019 Aug;69(8):1194-1198. PMID 31431779